CLINICAL TRIAL: NCT06829407
Title: Evaluation of the Effects of Different Methods Used in Subcutaneous Heparin Injections on Pain and Satisfaction
Brief Title: Effect of Different Subcutaneous Injection Methods on Pain and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ali Umit Yilmaz, Nurse, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TUTF-GOBAEK 202313|8
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pain, Acute; Injection Site
Keywords: pain; low molecular weight heparin; palm stimulator; extended injection time
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: this study is an experimental, parallel-group (intervention-control), randomized controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- injection time (Experimental): The application will be done by injecting for 30 seconds and then waiting for 10 seconds and ending the process.
  Interventions: Other: injection time
- palm stimulator (Experimental): By ensuring that the patient grasps the "palm stimulator" equipment in the palm during the injection and squeezes it in the palm throughout the injection. Tactile warning will be given. However, the injection process will last 10 seconds and the process will be terminated after waiting 10 seconds.
  Interventions: Other: palm stimulator
- injection time and palm stimulator (Experimental): Injection will be done for 30 seconds and then waited for 10 seconds and the process will be terminated, and the application will be done using equipment.
  Interventions: Other: injection time and palm stimulator
- control group (No Intervention): The injection process will last 10 seconds and the process will be terminated after waiting 10 seconds.

INTERVENTIONS:
Other: injection time — give an injection
  Arms: injection time
Other: palm stimulator — give an injection
  Arms: palm stimulator
Other: injection time and palm stimulator — give an injection
  Arms: injection time and palm stimulator

SUMMARY:
This study; In patients treated with subcutaneous heparin A randomized controlled trial was planned to determine the effect of the injection time and the device called "Palm Stimulator" to reduce the pain felt during injection.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* The one who is literate,
* No physical, mental disabilities or communication difficulties,
* Low Molecular Weight Heparin in the treatment plan,
* No history of allergy,
* Agreeing to participate in the research,
* There is no scar tissue, incision or infection in the area to be injected,
* Patients who will receive a 1-day injection and whose pain score is between 1-10 according to VAS will be admitted.

Exclusion Criteria:

* Who gave up participating in the research while continuing the research,
* Using subcutaneous insulin therapy,
* There is an amputation in the right/left arm area where the study will be performed,
* There is scar tissue, incision or signs of infection in the area to be injected,
* Patients who received injections for 1 day and whose pain score is 0 (zero) according to VAS will not be admitted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Scale Patient Identification Form | during injection procedure
  Patient Identification Form
  It was prepared by researchers by examining the literature on the subject. This form includes 5 questions that include some sociodemographic characteristics of the individual (age, gender, marital status, education status, employment status, etc.) and 8 questions that include characteristics related to health, illness and treatment (presence of chronic disease, body mass index, etc.).
Visual Scale for pain | during injection procedure
  Visual comparison scale for pain The scale consists of a single item, the scale is formed by a 10 cm long line on the horizontal plane. The leftmost side of the line (starting point) is scored as 0 (zero) and the rightmost side (ending point) is scored as 10 (ten) points for the highest possible pain. In order for the patient to score the pain, he/she is asked to mark a point on the line during the injection process. After marking, the distance from the starting point to the marked place is measured and the score is formed. The scale has been proven to be reliable in terms of Turkish as a result of the study conducted by Yaray et al.
Visual Comparison Scale for Satisfaction | during injection procedure
  Visual Comparison Scale for Satisfaction In this scale, scores between 0 and 10 were used to determine satisfaction levels. A score of 0 represented the least satisfaction level, while a score of 10 represented the highest satisfaction level. The Visual Analog Scale was used so that patients could express both their pain and satisfaction levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya Üniversitesi, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No